CLINICAL TRIAL: NCT04832698
Title: Survey of Current Interventional and Diagnostic Imaging Residents After Participation in Endovascular Simulator Training Regimen
Brief Title: Survey of Current Interventional and Diagnostic Imaging Residents After Participation in Endovascular Simulator Training
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0071; NCI-2020-06610 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0071 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-09-15; First posted 2021-04-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Malignant Vascular Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey administration): Participants complete a survey over 10 minutes before and after completing training and using the Mentice endovascular simulator device.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete survey

SUMMARY:
This study looks at the comfort of interventional and diagnostic imaging residents in performing simulated endovascular procedures after completing training on the Mentice endovascular simulator device. Implementation of a training curriculum with radiology residents interested in interventional radiology will help facilitate hands-on training in a low-risk environment and allow for safer future patient encounters.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To measure trainee comfort performing simulated endovascular procedures after completing training on the Mentice endovascular simulator device.

OUTLINE:

Participants complete a survey over 10 minutes before and after completing training and using the Mentice endovascular simulator device.

ELIGIBILITY:
Inclusion Criteria:

- Current interventional and diagnostic radiology residents participating in the training curriculum on the Mentice Endovascular Simulator will be eligible to participate in the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Current interventional and diagnostic radiology residents participating in the training curriculum on the Mentice Endovascular Simulator at MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Trainees' feelings about using simulation to help with procedural training | through study completion, an average of 1 year
  Will measure how trainees feel about using simulation to help with procedural training, and how comfortable trainees feel performing various endovascular procedures after undergoing training on the Mentice simulator machine.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Kuban, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org